CLINICAL TRIAL: NCT00162591
Title: Bispectral Index as an Analgesia Monitoring in Severely Ill Patient: Effect of Remifentanyl
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P040201 AT/AT/04-116
Record Dates: First submitted 2005-09-10; First posted 2005-09-13 (Estimated); Last update posted 2005-11-22 (Estimated); Status verified 2004-10

CONDITIONS: Pain
Keywords: Bispectral index; sedation; remifentanyl; Bronchoalveolar lavage; Intensive care; Nociceptive stimuli; Sedated patient; BIS variation
MeSH Terms: conditions — Pain | interventions — Remifentanil

INTERVENTIONS:
Drug: remifentanyl

SUMMARY:
The aim of this protocol is to study the prophylactic effect of remifentanil on bispectral index variation during a nociceptive stimuli.

DETAILED DESCRIPTION:
Pain is difficult to estimate in ICU because most of the patients are sedated. Bispectral index could be helpful in detecting this pain in ICU patients. Remifentanil is a morphinomimetic product with short half life that could be interesting for short nociceptive stimuli, as bronchoalveolar lavage.

The purpose of this study is to evaluate the impact of remifentanil infusion on bispectral index (BIS) variations during bronchoalveolar lavage.

It is a prospective, double blind study, versus placebo on 40 sedated and critically ill patients.

The hypothesis is that BIS can study analgesia in sedated patient.

ELIGIBILITY:
Inclusion Criteria:

* Sedated patient with mechanical ventilation with suspected nosocomial pneumonia

Exclusion Criteria:

* Pace maker
* Neurologic illness
* Hemodynamic instability
* Hypothermia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-10

PRIMARY OUTCOMES:
BIS variation during bronchoalveolar lavage

SECONDARY OUTCOMES:
Systolic blood pressure, diastolic blood pressure, heart rate viation

CONTACTS AND LOCATIONS:
Overall Officials: QUINTARD H Hervé, MD, Principal Investigator — Surgical ICU Bichat Claude Bernard (Paris, France)
Locations (1):
- Surgical ICU Bichat Claude Bernard, Paris, France

REFERENCES:
- [Derived] Quintard H, Pavlakovic I, Mantz J, Ichai C. Adjunctive remifentanil infusion in deeply sedated and paralyzed ICU patients during fiberoptic bronchoscopy procedure: a prospective, randomized, controlled study. Ann Intensive Care. 2012 Jul 16;2(1):29. doi: 10.1186/2110-5820-2-29. PMID 22800647